CLINICAL TRIAL: NCT04381455
Title: Evaluation of OSSIX® Bone in Maxillary Sinus Floor Augmentation
Brief Title: Evaluation of OSSIX® Bone in Sinus Elevation
Status: Completed | Type: Observational
Sponsor: Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo (Other)
Responsible Party: Principal Investigator, Luigi Canullo, Dr Luigi Canullo, DDS, Ph.D, Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo
Other Study IDs: DD-01
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Maxillary Sinus Floor Augmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: OSSIX Bone — subjects will be implanted with OSSIX Bone during sinus elevation surgery

SUMMARY:
A post marketing observational study to evaluate clinical performance of OSSIX Bone in maxillary sinus elevation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring vertical elevation of the maxillary sinus.
2. Residual alveolar bone height of edentulous maxilla below the floor of the maxillary sinus of > 4-5mm.
3. Males and females between 30-80 years old
4. Patients with healthy periodontal conditions (Treated periodontitis, PI<25%, BoP<25%)
5. Patients that are willing to sign an informed consent and participate in a clinical study
6. Generally fit and healthy and able to undergo oral surgical procedures under local anesthesia.
7. Teeth at the surgical site which required removal were extracted a minimum of 12 weeks prior to sinus floor elevation.

Exclusion Criteria:

1. Patients who smoke over 5 cigarettes/day
2. Pregnancy (confirmed by verbal inquiry)
3. Chronic systemic pathologies (e.g. diabetes) and neoplastic of the Oro-Facial District 4.
4. Patients taking bisphosphonates
5. Any sites where an implant already failed sites
6. Untreated Periodontitis
7. Dental sites with acute infections
8. Chronic inflammatory diseases of the oral cavity
9. Autoimmune diseases (cortisone intake)
10. Allergy declared to one or more medicaments to be used during treatment
11. Alcoholics patients and/or drug addicts
12. Patients with known collagen hypersensitivity.
13. Patients with sensitivity to porcine-derived materials.
14. History or malignant tumours of the maxillary sinus
15. History of local radiation therapy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that need sinus elevation
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Difference in Bone height from baseline | 1 year
Difference in bone volume | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Canullo, DDS, PhD, Principal Investigator — Study site
Locations (1):
- Studio Odont.Associato Dr.P.Cicchese E L.Canullo, Rome, Italy

IPD SHARING:
Plan to Share IPD: No